CLINICAL TRIAL: NCT01591980
Title: Effects of Perioperative Low-dose Pregabalin on Post-craniotomy Pain: A Two-centre Randomized Controlled Trial
Brief Title: Effects of Perioperative Pregabalin for Post-Craniotomy Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Pfizer Canada and the SMH ORA could not come into an agreement on responsibility to be the Importer of Record for the trial.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB-10-388
Record Dates: First submitted 2011-12-09; First posted 2012-05-04 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Postoperative Pain; Headache
Keywords: post-craniotomy pain; pregabalin; chronic post-craniotomy headache; Craniotomy
MeSH Terms: conditions — Pain, Postoperative; Headache | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pregabalin 100 mg (Experimental)
  Interventions: Drug: Pregabalin
- pregabalin 150 mg (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Sham Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Pre-operatively, one of the 2 doses of pregabalin (100 or 150 mg) or placebo will be given to patients 1 hour before the surgery. Post-operatively, patients will receive daily (split in 2 equal doses) pregabalin 100 mg, pregabalin 150 mg, or placebo for the first 14 post-operative days.
  Other Names: Lyrica
  Arms: Pregabalin 100 mg
Drug: pregabalin — Pre-operatively, one of the 2 doses of pregabalin (100 or 150 mg) or placebo will be given to patients 1 hour before the surgery. Post-operatively, patients will receive daily (split in 2 equal doses) pregabalin 100 mg, pregabalin 150 mg, or placebo for the first 14 post-operative days.
  Other Names: Lyrica
  Arms: pregabalin 150 mg
Drug: placebo — Identical placebo capsules will be administered in the same way.
  Other Names: Identical placebo capsules
  Arms: Placebo

SUMMARY:
Objective: To compare the incidence of chronic pain at 3 months among adults undergoing craniotomy between those received two different doses of pregabalin and those receiving placebo.

DETAILED DESCRIPTION:
Hypothesis: Perioperative pregabalin will reduce the incidence of chronic post-operative pain, and will reduce the opioid consumption, opioid-related side effects, and hospital length of stay compared with placebo in patients undergoing elective craniotomy.

Methods: 316 adults (18-65y), ASA I-III, undergoing elective craniotomy will be randomized to receive: 100mg or 150mg pregabalin or placebo once pre-operatively and 50mg or 75mg or placebo twice daily for 14 post-operative days. NRS pain scores, opioid consumption and side effects will be assessed up to 48h, and long-term pain at days 7, 14, 30, and 90. The primary analysis will involve the comparison between the 2 treatment groups together vs. placebo. A stepwise method will be used to evaluate the pairwise comparisons.

Outcomes: The primary outcome will be the incidence of chronic post-craniotomy pain at 3 mos. Important secondary outcomes are: neuropathic component of pain at 3 mos., total opioid consumption in the first 24h, and incidence and severity of opioid-related side effects at days 1, 2 and 7.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 to 65 years (limited to 65 years to lower the risk of over-sedation for elderly patients)
* Undergoing elective craniotomy (supratentorial or infratentorial) under general anaesthesia for: biopsy or resection of a tumour, clipping of an unruptured aneurysm, or excision of an arteriovenous malformation
* ASA physical status I-III

Exclusion Criteria:

* predicted need for prolonged post-operative ventilation (> 12 hours)
* chronic pain secondary to previous craniotomy
* known adverse reaction to drugs used (gabapentin, pregabalin, hydromorphone, and/or acetaminophen)
* prior use of pregabalin or gabapentin (within 2 weeks before surgery)
* current history of moderate to severe headaches (NRS ≥ 4) related to intracranial pathology (tumour pain) since it may be difficult to discriminate between ongoing tumour pain and surgery-related post-operative pain
* current history of migraines
* pre-existing chronic pain requiring chronic opioid use (30mg morphine equivalent within 4 weeks of surgery)
* currently taking any drug that could interact with pregabalin
* current history of alcohol or recreational drug abuse
* known or suspected addiction to narcotic substances or chronic narcotic use in the last 2 weeks
* history of malignant hyperthermia (contraindicates the anaesthesia protocol of this study)
* history of angioedema
* Body Mass Index ≤ 18.4 or ≥ 35
* history of untreated obstructive sleep apnea
* any condition that would contraindicate the use of patient-controlled analgesia (PCA)
* lacks fluency in English
* pre-existing renal impairment (for pregabalin elimination)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Chronic post-craniotomy pain | 3 months
  The primary outcome of this study will be the incidence of chronic post-craniotomy pain at 3 months

SECONDARY OUTCOMES:
neuropathic component of the pain at 3 months | 3 months
incidence of long-term pain at days 7 | Day 7
incidence of long-term pain at day 14 | Day 14
incidence of long-term pain at day 30 | Day 30
total opioid consumption in the first 24h | 24 hours
total patient-controlled analgesia (PCA)demands and delivered doses in 24h | 24 hours
post-operative pain scores at 24h | 24 hours
post-operative pain scores at 48h | 48 hours
incidence and severity of opioid-related side effects at day 2 | Day 2
incidence and severity of opioid-related side effects at Day 7 | Day 7
consumption of antiemetics in the first 24h | 24 hours
tracheal extubation time | within 24 hours
length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rigamonti, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada